CLINICAL TRIAL: NCT05867641
Title: VR&R: Providing Respite to Caregivers by Managing BPSDs and Improving QoL in People with Dementia Using Immersive VR-Therapy
Brief Title: VR&R: Providing Caregiver Respite by Managing BPSDs and Improving QoL in People with Dementia Using Immersive VR-Therapy
Acronym: VR&R
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Centre for Aging and Brain Health Innovation (Other); Ontario AHSC AFP Innovation Fund (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Lora Appel, Associate Professor, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VR&R
Record Dates: First submitted 2023-03-20; First posted 2023-05-22 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Dementia
Keywords: Non-pharmacological; Caregiver Respite; Virtual Reality; Home Based Care; Quality of Life; Behavioral and psychological symptoms of dementia; Mood; Well-Being; Serious Game
MeSH Terms: conditions — Dementia; Behavior | interventions — Smart Glasses; Oxymetholone

STUDY DESIGN:
Intervention Model Description: Pragmatic crossover interventional trial including a four-week home-based intervention (two weeks per condition) and two-week follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR&R Therapy - Solo First (Experimental): Recruited dyads will include one person diagnosed with dementia and their caregiver (e.g., family/friend). The caregiver will assist their loved ones with dementia to use VR-therapy at home. Caregivers may use the time while their loved ones are engaged for respite, remaining nearby to supervise and assist.
  For the first two weeks, only the caregiver will be present to use VR with the person with dementia. For the following two weeks, a research assistant will be present to use VR with the person with dementia.
  Interventions: Behavioral: Immersive VR Therapy in Head-Mounted Display (HMD) (Solo); Behavioral: Immersive VR Therapy in a Head-Mounted Display (HMD) (Social)
- VR&R Therapy - Social First (Experimental): Recruited dyads will include one person diagnosed with dementia and their caregiver (e.g., family/friend). The caregiver will assist their loved ones with dementia to use VR-therapy at home. Caregivers may use the time while their loved ones are engaged for respite, remaining nearby to supervise and assist.
  For the first two weeks, a research assistant will be present to use VR with the person with dementia. For the following two weeks, only the caregiver will be present.
  Interventions: Behavioral: Immersive VR Therapy in Head-Mounted Display (HMD) (Solo); Behavioral: Immersive VR Therapy in a Head-Mounted Display (HMD) (Social)

INTERVENTIONS:
Behavioral: Immersive VR Therapy in Head-Mounted Display (HMD) (Solo) — Caregivers will be trained to administer VR&R therapy to their loved ones with dementia, in their private home/residence. Participants with dementia will view immersive VR experiences using a commercially-available VR head-mounted device for up to 30 minutes a time, approximately every other day (or as desired), for two weeks. The caregiver will use the custom application on a tablet to select and monitor what their loved one sees in VR.
  Staying nearby to monitor for safety and assistance, the caregiver may choose to use the time when their loved one is engaged to take some respite time for themselves (e.g., make a cup of coffee, have an uninterrupted phone call).
  Other Names: Solo VR Therapy
Behavioral: Immersive VR Therapy in a Head-Mounted Display (HMD) (Social) — Participants with dementia will view immersive VR experiences using a commercially-available VR head-mounted device for up to 30 minutes a time, 2 to 3 times per week, for 2 weeks. A research assistant who is trained in dementia care will use the custom application on a tablet to select and monitor what their loved one sees in VR.
  Staying nearby to monitor for safety and assistance, the caregiver may choose to use the time when their loved one is engaged to take some respite time for themselves (e.g., make a cup of coffee, have an uninterrupted phone call).
  Other Names: Social VR Therapy

SUMMARY:
The goal of this interventional trial is to learn about how immersive Virtual Reality (VR) therapy can be used at home by individuals with dementia, with assistance from their informal (e.g., friend/family) caregivers.

The main question it aims to answer are:

1. Can caregivers receive quality respite time by using VR-therapy at home with their loved ones with dementia? Does this intervention reduce feelings of burden and improve well-being and resilience for caregivers?
2. Does VR-therapy help to manage behavioural and psychological symptoms (e.g., mood, apathy, agitation) and improve quality of life for individuals with dementia?
3. What types of VR "medium" (passive or cooperative) are most effective for achieving the above objectives?

Participant pairs will be asked to:

* Take part in an initial at-home VR technology training session and complete a series of brief questionnaires (e.g., health history/technology use, well-being/quality of life, symptoms of dementia)
* Use "VR&R" (VR Rest & Relaxation Therapy) for a period of 4 weeks (30 minute sessions, desired frequency), and answer a brief set of questions after each VR&R session
* Provide feedback on the VR&R intervention in semi-structured interview with the researcher and answer additional questionnaires at a 2-week follow-up

During VR&R sessions, participants with dementia will have the opportunity to choose to watch (1) immersive 360-degree videos (e.g., of a live performance, or beach) on their own and (2) experience the same VR videos together with a researcher.

Caregivers will be asked to assist their loved one with dementia to use VR&R by helping to put on the VR headset, selecting a VR experience through a user-friendly application, and remaining nearby to supervise and provide assistance as needed. During VR&R sessions, caregivers may use this time to take a personal break or complete short tasks (e.g., make a cup of coffee, have an uninterrupted phone call).

DETAILED DESCRIPTION:
Caregivers of individuals with dementia experience twice as much distress as those providing care for other seniors. This burden is particularly common when the person with dementia displays aggression. A number of recent studies have indicated that Virtual Reality (VR)-therapy is a safe, acceptable, and enjoyable non-pharmacological intervention for individuals with dementia, with potential to manage symptoms and promote quality of life. However, further research is needed to determine how to best design VR-therapy for this purpose. Moreover, it is not yet known whether VR is helpful for providing respite for caregivers. In this study, the investigators aim to determine whether "VR&R", an immersive VR-therapy, is helpful for providing caregiver respite and managing symptoms of dementia (mood, apathy, agitation). Additionally, this study will explore what type of VR "medium" is most effective for achieving these outcomes. The VR&R intervention includes a user-friendly web-application that caregivers can use to select among three different multi-sensory mediums for their loved one with dementia to experience (1) "Solo VR": 360-degree videos that simulate real-life environments (the ocean, watching a ballet) and (2) "Social VR": where a researcher interacts with the participants while using VR. Participants will use VR&R at home for up to 30 minutes at a time, for four weeks. Outcomes will be evaluated using mixed methods (questionnaires, semi-structured interviews, observations, objective metrics of VR usage). The investigators predict that the intervention will provide caregivers with uninterrupted time to complete brief tasks that they may not have been able to otherwise, improving well-being and reducing feelings of burden. This study's findings will have implications for designing and implementing home-based VR interventions, including which types of VR experiences keep individuals with dementia engaged the longest, are easiest to use, and are seen as most beneficial by end-users.

ELIGIBILITY:
Inclusion Criteria: People with dementia

* Individuals who are 65 years of age or older
* Individuals living at home with a family caregiver
* Individuals diagnosed with dementia

Exclusion Criteria:

* Individuals with open wounds on face (sutured lacerations exempted)
* Individuals with a history of seizures or epilepsy
* Individuals with a pacemaker
* Individuals with head trauma or stroke leading to their current admission
* Individuals with cervical conditions or injuries that would make it unsafe for them to use the VR headset
* Individuals who identify as being legally blind
* Individuals with alcohol related dementia/ Korsakoff syndrome.
* Individuals who have a Public Guardian and Trustee (PGT) as Substitute Decision Maker (SDM)
* Individuals who cannot speak and understand English

Caregiver inclusion criteria:

* Individuals who identify as a primary caregiver for the PwD
* Individuals who have access to the internet through a device (computer, tablet, or mobile phone) that can be used during the study

Caregiver exclusion criteria:

* Individuals who cannot speak and understand English
* Individuals who are cognitively unable to provide informed consent for themselves
* Identify as legally blind

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Caregiver Respite and Burden | 6 Weeks
  Unpaid Caregivers: Short Zarit Burden Interview The Short Zarit Burden Interview tool will be completed by caregiver-participants and will be used to evaluate subjective feelings of caregiver burden associated with being a caregiver for the person with dementia. The Short Zarit Burden Interview is a 6-item questionnaire that employs a 5-point Likert scale. Total scores range from 0-24 where higher scores indicate greater feelings of caregiver burden.
  Paid Caregivers: Professional Care Team Burden Scale The 10-item Professional Care Team Burden (PCTB) Scale is a validated tool designed to assess the burden experienced by professional caregivers working in dementia care settings such as nursing homes. It evaluates three dimensions of burden: subjective burden (individual emotional strain), organizational burden (workplace factors), and structural burden (systemic or institutional challenges).
Change in Caregiver Respite and Burden: Caregiver Phone Interview | 6 Weeks
  The caregiver will be asked to take part in a pre- and post- intervention phone interview (approximately 15 minutes in length, audio-recorded). The interview will include open-ended questions to gather qualitative information on the impact of the VR intervention on the caregiver and PwD (i.e., whether there were any changes to baseline PwD & caregiver well-being/QoL, BPSD, caregiver burden, and caregiver respite following the intervention), as well as feedback on the VR mediums in terms of their ability to promote caregiver respite.
Change Caregiver Well-Being | 6 Weeks
  WHO-5 Well-Being Index will be administered to caregiver-participants to evaluate subjective wellbeing. The WHO (Five) is a 5-item questionnaire employing 6-point Likert scales. Calculated scores range from 0-25. A score of 0 represents the worst possible and a score of 25 represents the best possible quality of life. A score below 13 represents poor wellbeing. A change of 10% represents a significant change in wellbeing.
Change in Caregiver Respite and Burden: Post-Session Log | 4 Weeks
  Caregivers will be asked to describe their time while the PwD was using VR in a paper-based log. This tool aims to capture if the caregiver was able to obtain additional respite, and the degree to which they were able to obtain respite (i.e., the degree to which caregivers were able to remain vigilant and at the same time detach and focus on their own task). Caregivers will also have the opportunity to record observations of the PwD's reactions to/experience with the VR intervention, as well as additional feedback and reflections of their own or from discussion with the PwD.
Change in Caregiver Resilience | 6 Weeks
  The 10-item Connor-Davidson Resilience Scale (CD-RISC) is a condensed version of the original 25-item scale, designed to efficiently measure resilience, the ability to adapt and thrive in the face of adversity. Each of its 10 items is rated on a 5-point Likert scale, with higher scores indicating greater resilience. The scale emphasizes key resilience traits such as adaptability, persistence, and emotional regulation. Validated across diverse populations, it has shown strong reliability, internal consistency, and construct validity. Its brevity and ease of use make it a valuable tool for both research and clinical settings, especially when time is limited.

SECONDARY OUTCOMES:
Change in PwD Behavioural and Psychological Symptoms of Dementia: Neuropsychiatric Symptoms | 6 Weeks
  The Neuropsychiatric Inventory-Questionnaire (NPI-Q) will be completed by the caregiver. The NPI-Q is a 12-item questionnaire that measures neuropsychiatric symptoms (e.g., related to related to mood, behavioural disturbance) as well as caregiver distress corresponding to reported symptoms.
Immediate Impact of Intervention on PwD Mood | 4 Weeks
  Participants with dementia will be prompted to select from a set of eight faces displaying different emotions, immediately before and after each VR-therapy session. These include positive emotions (happy, joyful, relaxed) and negative emotions (anxious, sad, angry, confused, indifferent). These metrics will be collected before and after each intervention session (i.e., at a time-interval of approximately 30 minutes, depending on session length.)

OTHER OUTCOMES:
Usability/Preference: System Usability Scale (SUS) | 6 Weeks
  The System Usability Scale (SUS) will be completed by the caregiver to evaluate device usability/ease-of-use of the VR intervention (head-mounted device and VR&R application) used during the study. The SUS is a 10-item questionnaire employing 5-point Likert scales. Calculated scores range from 0-100. Higher scores indicate better system usability.
Usability/Preference: Semi-Structured Interviews | 6 Weeks
  The caregiver will take part in a semi-structured interview post-intervention. The interview will include open-ended questions to explore the acceptability and usability the 2 different VR-mediums, including suggestions for improvement.
PwD Simulator Sickness | Baseline
  During the initial home training (pre-intervention), the researcher will observe the participant's reactions to a brief "neutral" VR video (a nature scene). The researcher will then administer the Fast Motion Sickness Scale (FMS). The scale asks the participant to rate any feelings of motion sickness on a scale of 0 to 20 where 0 indicates no motion sickness and 20 indicates a great deal of motion sickness (on the brink of vomiting). Participants with a score of 15 or higher will be withdrawn from the study.
PwD Preferences/Reactions to VR: Post-Session Experience Ratings | 4 Weeks
  Immediately after each session, participants with dementia will be prompted to rate their experience on a visual analog "Star" scale (range of 1 to 5), where 1 indicates the worst possible experience and 5 indicates the best possible experience.
PwD Preferences/Reactions to VR: Post Session Log | 4 Weeks
  Caregivers will be asked to record any observations and feedback related to their their loved one's reactions to VR (e.g., enjoyment, relaxation, engagement, anxiety/apprehension; what did/did not go well). Caregivers will be asked to make these recordings immediately after intervention sessions.
PwD Preferences/Reactions to VR: Time Spent in Each VR Medium | 4 Weeks
  This objective metrics of VR usage will be will be unobtrusively collected through the VR&R application for the duration of the study.
PwD Preferences/Reactions to VR: Head Movements in VR | 4 Weeks
  This objective metrics of VR usage will be will be unobtrusively collected through the VR&R application for the duration of the study.
Cognition (Participant with Dementia) | Baseline
  The Mini Mental State Exam (MMSE) will be administered to the PwD at baseline. This is a widely used cognitive screening test consisting of 12 questions administered orally. Scores range from 0-30, with scores of 0-9 suggesting severe cognitive impairment/late stage dementia, scores of 10-19 suggesting moderate cognitive impairment/middle stage dementia, scores of 20-25 suggesting mild cognitive impairment/early stage dementia, and scores of 26-30 suggesting possibly normal cognition.
Gender Expression (Caregiver) | Baseline
  A short form of the Personality Attributes Questionnaire with 8 items (PAQ-8) used to assess femininity and masculinity, which has been found to be a valid screening measure to assess gender expression. Scores on each scale are range from 0-32. On the masculine and masculine-feminine subscales, higher scores indicate a greater level of masculinity. On the feminine subscale, a higher score indicates a greater level of femininity.

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (7):
  - Acclaim Health, Oakville, Ontario
  - Chester Village, Toronto, Ontario
  - Circle of Care, Toronto, Ontario
  - Toronto Grace Hospital - Main Site, Toronto, Ontario
  - Toronto Grace Hospital - Remote Care Monitoring, Toronto, Ontario
  - Toronto Grace Hospital - Specialized Care Centre, Toronto, Ontario
  - McGill Dementia Education Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson-Hanley C, Arciero PJ, Brickman AM, Nimon JP, Okuma N, Westen SC, Merz ME, Pence BD, Woods JA, Kramer AF, Zimmerman EA. Exergaming and older adult cognition: a cluster randomized clinical trial. Am J Prev Med. 2012 Feb;42(2):109-19. doi: 10.1016/j.amepre.2011.10.016. PMID 22261206
- [Background] Appel L, Appel E, Bogler O, Wiseman M, Cohen L, Ein N, Abrams HB, Campos JL. Older Adults With Cognitive and/or Physical Impairments Can Benefit From Immersive Virtual Reality Experiences: A Feasibility Study. Front Med (Lausanne). 2020 Jan 15;6:329. doi: 10.3389/fmed.2019.00329. eCollection 2019. PMID 32010701
- [Background] Appel L, Kisonas E, Appel E, Klein J, Bartlett D, Rosenberg J, Smith C. Introducing virtual reality therapy for inpatients with dementia admitted to an acute care hospital: learnings from a pilot to pave the way to a randomized controlled trial. Pilot Feasibility Stud. 2020 Oct 31;6(1):166. doi: 10.1186/s40814-020-00708-9. PMID 33292729
- [Background] Appel L, Kisonas E, Appel E, Klein J, Bartlett D, Rosenberg J, Smith CN. Administering Virtual Reality Therapy to Manage Behavioral and Psychological Symptoms in Patients With Dementia Admitted to an Acute Care Hospital: Results of a Pilot Study. JMIR Form Res. 2021 Feb 3;5(2):e22406. doi: 10.2196/22406. PMID 33533720
- [Background] Appel L, Ali S, Narag T, Mozeson K, Pasat Z, Orchanian-Cheff A, Campos JL. Virtual reality to promote wellbeing in persons with dementia: A scoping review. J Rehabil Assist Technol Eng. 2021 Dec 21;8:20556683211053952. doi: 10.1177/20556683211053952. eCollection 2021 Jan-Dec. PMID 35024166
- [Background] Baker JR, Webster L, Lynn N, Rogers J, Belcher J. Intergenerational Programs May Be Especially Engaging for Aged Care Residents With Cognitive Impairment: Findings From the Avondale Intergenerational Design Challenge. Am J Alzheimers Dis Other Demen. 2017 Jun;32(4):213-221. doi: 10.1177/1533317517703477. PMID 28506126
- [Background] D'Cunha NM, Nguyen D, Naumovski N, McKune AJ, Kellett J, Georgousopoulou EN, Frost J, Isbel S. A Mini-Review of Virtual Reality-Based Interventions to Promote Well-Being for People Living with Dementia and Mild Cognitive Impairment. Gerontology. 2019;65(4):430-440. doi: 10.1159/000500040. Epub 2019 May 20. PMID 31108489
- [Background] Dermody G, Whitehead L, Wilson G, Glass C. The Role of Virtual Reality in Improving Health Outcomes for Community-Dwelling Older Adults: Systematic Review. J Med Internet Res. 2020 Jun 1;22(6):e17331. doi: 10.2196/17331. PMID 32478662
- [Background] Huygelier H, Schraepen B, van Ee R, Vanden Abeele V, Gillebert CR. Acceptance of immersive head-mounted virtual reality in older adults. Sci Rep. 2019 Mar 14;9(1):4519. doi: 10.1038/s41598-019-41200-6. PMID 30872760
- [Background] Munoz J, Mehrabi S, Li Y, Basharat A, Middleton LE, Cao S, Barnett-Cowan M, Boger J. Immersive Virtual Reality Exergames for Persons Living With Dementia: User-Centered Design Study as a Multistakeholder Team During the COVID-19 Pandemic. JMIR Serious Games. 2022 Jan 19;10(1):e29987. doi: 10.2196/29987. PMID 35044320
- See also: VR&R Project Website — https://www.prescribingvr.com/vrnr